CLINICAL TRIAL: NCT07024407
Title: Phase 1b Study of Andecaliximab in Participants With Spinal Cord Injury at Risk of Developing Heterotopic Ossification
Brief Title: A Study of Andecaliximab in People With Spinal Cord Injury at Risk for Bone Growth Outside of the Normal Skeleton.
Acronym: ANDECA-HO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ashibio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ASH-HO-201
Record Dates: First submitted 2025-05-20; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Heterotopic Ossification (HO)
Keywords: Heterotopic Ossification; traumatic spinal cord injury
MeSH Terms: conditions — Ossification, Heterotopic | interventions — andecaliximab

STUDY DESIGN:
Intervention Model Description: All participants will receive andecaliximab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Andecaliximab (Experimental): All participants will receive andecaliximab whether at risk for developing HO or at risk for worsening of early HO.
  Interventions: Drug: Andecaliximab

INTERVENTIONS:
Drug: Andecaliximab — Participants will receive weekly subcutaneous injections of andecaliximab during inpatient hospitalization, clinic visit, or self-administration if discharged from the hospital

SUMMARY:
This is an open-label study of andecaliximab in participants at risk of developing bone where bone should not be, such as in muscle, tendons, and other soft tissues following traumatic spinal cord injury. The goal of this study is to assess the safety of andecaliximab, how much drug is in the body over time (pharmacokinetics/PK), and how it affects the body (pharmacodynamics/PD) in participants who have had a recent traumatic spinal cord injury.

DETAILED DESCRIPTION:
Safety: To evaluate the safety profile of andecaliximab in participants with spinal cord injurySCI at risk for Heterotopic Ossification.

PK: To describe the PK profile of andecaliximab in all participants.

Secondary Objective:

PD: To describe the PD profile of andecaliximab in all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 89 years.
2. History of traumatic SCI that occurred a minimum of 10 days prior to first study dose.
3. No significant HO identified by CT as defined in the Imaging Charter and meeting one of the following sets of criteria based on TPBS at end of screening:

The Inflammatory Group: Inflammation consistent with developing HO The Early HO Group: The third phase on TPBS shows minimal extraskeletal uptake

The Prophylactic High-Risk Group: No findings consistent with increased risk of HO but meets all of the following clinical risk factors for HO:

1. Within 1 month of injury AND
2. AIS Grade A AND
3. Male AND
4. Age 18 to 45 years 4. Participant or legal representative able and willing to give informed consent and to adhere to the visits schedule and study procedures.

5. Able to understand, undergo, and perform all protocol related procedures. 6. Agrees to provide access to all relevant current and historical medical records

Exclusion Criteria:

1. History of:

   1. Known monogenic disorder associated with HO.
   2. Bone or mineral disorder unrelated to HO or SCI.
   3. Malignancy (within the past 5 years). Untreated active infection at the time of enrollment Uncontrolled hypoparathyroidism or hyperparathyroidism Uncontrolled hyperthyroidism, based on participant report or chart review. Hyperthyroidism is defined by the presence of both a TSH level below the normal range and elevated T4.
   4. Current infection with COVID-19 or COVID-19 infection within 1 month of Study Day 1 if treated with nirmatrelvir/ritonavir or other COVID-19 antiviral with a risk of rebound. (If a potential participant is experiencing mild COVID-19-like symptoms, they should wait until they are asymptomatic and/or rule out COVID-19 infection by local COVID-19 PCR testing prior to on-site screening.) Asymptomatic patients are not required to undergo COVID-19 testing.
   5. COVID-19 vaccine within 1 month of Study Day 1.
2. Use of the following medication:

   1. Current or chronic use of tetracycline drugs
   2. Activated (1,25-OH) vitamin D (vitamin D2 and D3 allowed), phosphate or calcium supplements within 1 week of Study Day 1
   3. Treatment with another investigational product within 5 half lives of last dose at the time of Study Day 1 or one month, whichever is longer.
3. History of allergy or hypersensitivity to andecaliximab or its excipients.
4. Any of the following abnormalities detected on laboratory evaluation prior to Study Day 1:

   1. 25-OH vitamin D <16 ng/mL (<39.94 nmol/L).
   2. Current albumin corrected serum calcium level <8.0 mg/dL or >11 mg/dL, or requiring treatment with IV fluids and/or bisphosphonates for hypercalcemia at time of enrollment.
   3. Impaired renal function. (estimated glomerular filtration rate [eGFR] < 40 mL/min/1.73m2)
   4. Hepatic panel [aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, direct bilirubin, lactate dehydrogenase (LDH)] >3 × ULN for ageHemoglobin <9.5 g/dL (<5.9 mmol/L).
   5. Absolute neutrophil count (ANC) <1,500 mm3(<1.5 × 109/L).
   6. Platelets <75,000/μL (<75 × 109/L).
5. Breastfeeding.
6. Pregnancy, planned pregnancy, or unwillingness to use acceptable birth control during the study and for 90 days after the last dose.
7. Simultaneous participation in another interventional clinical trial.
8. Any other significant medical condition or disability or biochemical or hematologic abnormalities, that in the opinion of the Investigator would expose the participant to undue risk, prevent the conduct of study procedures, or confound the study results.
9. Employees of the Sponsor, study site, or CRO involved in the conduct of the study or immediate family members thereof.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of andecaliximab in participants with SCI at risk for HO | From signing of the informed consent form until the end of the Safety Follow-up Period (4 weeks after week 9 or Early Termination)
  Incidence and severity of all serious adverse events (SAEs) and all treatment-emergent adverse events (TEAEs)
To describe the PK profile of andecaliximab in all participants | From baseline (Week 1) through Week 9 or Early Termination
  PK parameters (area under the time-concentration curve [AUC], maximum concentration [Cmax],
To describe the PK profile of andecaliximab in all participants | From baseline (Week 1) through Week 9 or Early Termination
  PK concentration at steady state [Ctrough]) describing the profile of andecaliximab

SECONDARY OUTCOMES:
To describe the PD profile of andecaliximab in all participants | From baseline (Week 1) through Week 9 or Early Termination
  Andecaliximab MMP9 target coverage in plasma over time

OTHER OUTCOMES:
Exploratory: To evaluate the efficacy of andecaliximab to inhibit new HO or continued development of HO in all participants | From baseline (Week 1) to Week 9
  Radiographic studies to determine percent of participants with new HO lesion; and percent of participants with critical new HO volume
To evaluate the response to adecaliximab in participant function | From baseline (Week 1) to Week 9
  Changes in passive range of motion testing (PROM)/active range of motion testing (AROM)
To evaluate the response to adecaliximab in participant function | From baseline (Week 1) to Week 9
  Changes in International Standard for Neurological Classification of Spinal Cord Injury (ISNCSCI)
To evaluate the response to andecaliximab in participant pain | From baseline (Week 1) to Week 9
  Changes in International Spinal Cord Society (ISCOS) Spinal Cord Injury Pain Classification

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Park, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Denver, Colorado, United States